CLINICAL TRIAL: NCT00844428
Title: An Open-Label, Multi-Center Controlled Clinical Trial Of Eculizumab in Adolescent Patients With Plasma Therapy-Sensitive Atypical Hemolytic Uremic Syndrome (AHUS)
Brief Title: Open Label Controlled Trial of Eculizumab in Adolescent Patients With Plasma Therapy-Sensitive aHUS
Acronym: aHUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C08-003B; BB-IND 11075; EudraCT Number 2008-006955-28
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Atypical Hemolytic Uremic Syndrome
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eculizumab (Experimental)
  Interventions: Drug: eculizumab

INTERVENTIONS:
Drug: eculizumab — All patients received open-label eculizumab administered intravenously on the following dose schedule: Induction dose - 900 mg per week for four weeks and a dose of 1200 mg one week later; Maintenance dose - 1200 mg every two weeks. Patients who received plasma exchange or infusion during the eculizumab treatment period received a supplemental dose of 600 mg within one hour before plasma infusion or within one hour after the completion of each plasma exchange.

SUMMARY:
The purpose of this study is to determine whether eculizumab is safe and effective in the treatment of adolescent patients with plasma therapy-sensitive Atypical Hemolytic-Uremic Syndrome (aHUS).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between ages from 12 and up to 18 years of age weighing ≥ 40 kg who have been diagnosed with Atypical Hemolytic-Uremic Syndrome (aHUS).
2. Patients must be receiving PT for aHUS and must be observed to receive ≥ 1 PT treatment every two weeks and no more than 3 PT treatments/week (at an unchanged frequency) for at least 8 weeks before the first dose of IP.
3. Platelet Count Pre-PT Baseline Set-Point (collected in the hours before the Qualifying PT Episode) is within 75% of the average of the pre-PT platelet counts collected at Screening and during the Observation Period.
4. Known complement regulatory protein genetic abnormality.
5. Lactate dehydrogenase (LDH) level at screening or at the onset of the current aHUS episode was ≥ ULN. If LDH is normal at screening, other markers indicative of ongoing hemolysis such as haptoglobin, schistocytes should be evaluated and discussed with Sponsor.
6. Creatinine level ≥ ULN for age.
7. Female patients of childbearing potential must be practicing an effective, reliable and medically approved contraceptive regimen during the entire duration of the study, including the follow-up period and for up to 5 months following eculizumab treatment discontinuation.
8. Patient's parents/legal guardian must be willing and able to give written informed consent and patient must be willing to give written informed assent (if applicable as determined by the IRB/IEC).
9. Able and willing to comply with study procedures.

Exclusion Criteria:

1. TTP, (defined as ADAMTS-13 activity <5%) from an historical observation (prior to initiation of plasma therapy) or as tested at the screening visit by the central laboratory.
2. Malignancy within 5 years of screening.
3. Typical HUS (Shiga toxin +).
4. Known HIV infection.
5. Identified drug exposure-related HUS.
6. Infection-related HUS.
7. HUS related to bone marrow transplant.
8. HUS related to vitamin B12 deficiency.
9. Patients with a confirmed diagnosis of sepsis.
10. Presence or suspicion of active and untreated systemic bacterial infection that, in the opinion of the Investigator confounds an accurate diagnosis of aHUS or impedes the ability to manage the aHUS disease.
11. Pregnancy or lactation.
12. Unresolved meningococcal disease.
13. Known Systemic Lupus Erythematosus (SLE) or antiphospholipid antibody positivity or syndrome.
14. Any medical or psychological condition that, in the opinion of the investigator, could increase the patient's risk by participating in the study or confound the outcome of the study.
15. Patients who have received previous treatment with eculizumab.
16. Patients receiving IVIg within 8 weeks or Rituximab therapy within 12 weeks of the screening visit.
17. Patients receiving other immunosuppressive therapies such as steroids, mTOR inhibitors or tacrolimus are excluded unless: [1] part of an established post-transplant anti-rejection regime, [2] patient has confirmed anti-CFH antibody requiring immunosuppressive therapy, and [3] dose of such medications have been unchanged for at least 4 weeks prior to the screening period and throughout the Obeservation Period or [4] patient is experiencing an acute aHUS relapse immediately after transplant.
18. Patients receiving Erythrocyte Stimulating Agents (ESAs) unless already on a stable dose for at least 4 weeks prior to the screening period or a washout period of at least 2 weeks from the last dose of ESA therapy.
19. Participation in any other investigational drug trial or exposure to other investigational agent, device, or procedures beginning 4 weeks prior to screening and throughout the entire trial.
20. Hypersensitivity to eculizumab, to murine proteins, or to one of the excipients.
21. Patients between the ages from 12 and up to 18 years weighing < 40 kg.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Toronto, Canada
- France (6):
  - Bois-Guillaume
  - Bordeaux
  - Lyon
  - Nantes
  - Paris
  - Starsbourg
- Hanover, Germany
- Genova, Italy
- Nijmegen, Netherlands
- Stockholm, Sweden
- United Kingdom (2):
  - Exeter
  - Glasgow

REFERENCES:
- [Derived] Pugh D, O'Sullivan ED, Duthie FA, Masson P, Kavanagh D. Interventions for atypical haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Mar 23;3(3):CD012862. doi: 10.1002/14651858.CD012862.pub2. PMID 33783815
- [Derived] Legendre CM, Licht C, Muus P, Greenbaum LA, Babu S, Bedrosian C, Bingham C, Cohen DJ, Delmas Y, Douglas K, Eitner F, Feldkamp T, Fouque D, Furman RR, Gaber O, Herthelius M, Hourmant M, Karpman D, Lebranchu Y, Mariat C, Menne J, Moulin B, Nurnberger J, Ogawa M, Remuzzi G, Richard T, Sberro-Soussan R, Severino B, Sheerin NS, Trivelli A, Zimmerhackl LB, Goodship T, Loirat C. Terminal complement inhibitor eculizumab in atypical hemolytic-uremic syndrome. N Engl J Med. 2013 Jun 6;368(23):2169-81. doi: 10.1056/NEJMoa1208981. PMID 23738544

RESULTS

PARTICIPANT FLOW:
Recruitment Details: C08-003A/B combined 2 studies: one for adults (C08-003A, N=15) and one for adolescents (C08-003B, N=5) Please refer to NCT008838513 for combined studies with enrollment number corresponding to each individual study
Pre-assignment Details: Patients receiving PT for aHUS and observed to receive ≥ 1 PT every two weeks, and no more than 3 PT treatments/week for at least 8 weeks before the first dose of eculizumab. Patients who met the eligibility criteria during the Observation Period were enrolled into the Treatment Period which commenced with the first eculizumab dose.
Period: Screening Period
Arm/Group | Eculizumab
Started | 23
Completed | 20
Not Completed | 3
Not completed — Screen Failure | 3
Period: Observation Period (8 Weeks)
Arm/Group | Eculizumab
Started | 20
Completed | 20
Not Completed | 0
Period: Treatment Period (26 Weeks)
Arm/Group | Eculizumab
Started | 20
Completed | 20
Not Completed | 0
Period: Extension Treatment Period
Arm/Group | Eculizumab
Started | 19
Completed | 18
Not Completed | 1
Not completed — Death | 1
Period: Post Treatment Period (Patients Who Disc
Arm/Group | Eculizumab
Started | 5
Completed | 4
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all patients who received any amount of eculizumab, and were considered evaluable for safety and efficacy analyses. For both the efficacy and safety analyses, all 20 patients who were treated with study drug were included in the ITT population.
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.3 (14.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With TMA Event-free Status
Description: TMA Event-free status is defined as the absence for at least 12 weeks of [1] decrease in platelet count of > 25% from the Platelet Count Pre-PT Baseline Set Point; [2] PT while the patient is receiving eculizumab, and [3] new dialysis.
Time Frame: Through 26 weeks
Population: The tabulations of the proportions of patients who achieved a TMA Event-Free status through 26 weeks were performed for the ITT population. Exact binomial 95% confidence intervals were produced for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Percentage of Participants | 80 [56 to 94]
Statistical Analysis 1: Comparison: Eculizumab; With a total of 20 patients enrolled between both protocols and, assuming that the true expected probability of TMA Event-Free for eculizumab-treated patients is 40%, then the study had 93.5% power to detect a statistically significant difference. Up to approximately 30 patients were to be enrolled. All analyses were based on the pooled data from the two protocols: C08-003A (adult) and C08-003B (adolescent), a similar protocol, for patients <18 years with aHUS; Test type: Superiority or Other; Percent of TMA event-free responders = 80, 95% CI 2-sided [56 to 94]

2. Primary Outcome: Percentage of Patients With Hematologic Normalization
Description: Hematologic Normalization was defined as normalization of both platelet count and lactic dehydrogenase (LDH) sustained for at least two consecutive measurements which spanned a period of at least four weeks.
Time Frame: Through 26 weeks
Population: Tabulations of the proportion of patients who achieved a hematologic normalization through 26 weeks were performed for the ITT population. Exact binomial 95% confidence intervals were produced for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Percentage of Participants | 90 [68 to 99]
Statistical Analysis 1: Comparison: Eculizumab; All analyses were based on the pooled data from the two protocols: C08-003A (adult) and C08-003B (adolescent), a similar protocol, for patients <18 years with aHUS; Test type: Superiority or Other; Percent of hematologic normalization = 90, 95% CI 2-sided [68 to 99]

3. Primary Outcome: Percentage of Patients With Complete TMA Response
Description: The proportion of patients who achieved a Complete TMA Response from baseline through 26 weeks of treatment with eculizumab was determined. Complete TMA Response was defined as Hematologic Normalization plus improvement in renal function (defined as (≥25% reduction from baseline in serum creatinine), which was sustained for two consecutive measurements over a period of at least four weeks.
Time Frame: Through 26 weeks
Population: Tabulations of the proportion of patients who achieved a complete TMA response from baseline through 26 weeks were performed. For this endpoint, for any relevant proportions, exact binomial 95% confidence intervals were produced.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Percentage of Participants | 25 [9 to 49]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Percent of complete TMA response = 25, 95% CI 2-sided [9 to 49]

4. Secondary Outcome: TMA Intervention Rate
Description: TMA Intervention Rate (# PE/PI and # Dialysis Events/Patient/Day) in the eculizumab treatment period (from baseline through 26 weeks) for PE/PI and (from the fifteenth day following the first eculizumab dose through 26 weeks) for new dialysis events was compared with the TMA Intervention Rate during the pre-eculizumab treatment period.
Time Frame: Through 26 weeks
Population: A signed rank test assessed differences in magnitudes of change in TMA intervention rate between the pre-eculizumab treatment period and during eculizumab treatment period for ITT population.
Measure: Mean (Standard Deviation); unit: #events/patient/day
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
#events/patient/day | 0 (0)
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.29

5. Secondary Outcome: Platelet Count Change From Baseline to 26 Weeks
Time Frame: From Baseline to 26 Weeks
Population: Change from baseline platelet counts were analyzed for the ITT population using a repeated measurement ANOVA model. A least squares (LS) mean for the change from baseline was produced for each study day for which a measurement of platelet count was scheduled. Significance of change was assessed at the 5% level at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
10^9 cells/L | 6.75 [-15.73 to 29.23]
Statistical Analysis 1: Comparison: Eculizumab; All analyses were based on the pooled data from the two protocols: C08-003A (adult) and C08-003B (adolescent), a similar protocol, for patients <18 years; Test type: Superiority or Other; p = 0.5423, ANOVA; Change from baseline were analyzed using a repeated measurement ANOVA model with time and baseline as fixed effects and subject as a random effect; LS mean change from baseline = 6.75, 95% CI 2-sided [-15.73 to 29.23]

6. Secondary Outcome: Percentage of Patients With Platelet Count Normalization
Description: Platelet count normalization was defined as the platelet count observed to be ≥150 x 10^9/L on at least two consecutive measurements which span a period of at least four weeks
Time Frame: Through 26 Weeks
Population: The tabulations of the proportion of patients who achieved platelet count normalization through 26 weeks were performed for the ITT population. Exact binomial 95% confidence intervals were produced for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Percentage of Participants | 90 [68 to 99]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Percent of platelet count normalization = 90, 95% CI 2-sided [68 to 99]

7. Secondary Outcome: Percentage of Patients With TMA Event-free Status
Description: as for outcome 1
Time Frame: Through End of Study, Median Exposure 156 Weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Percentage of Participants | 95 [75 to 100]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Percent of TMA event-free responders = 95, 95% CI 2-sided [75 to 100]

8. Secondary Outcome: Percentage of Patients With Hematologic Normalization
Description: as for outcome 2
Time Frame: Through End of Study, Median Exposure 156 Weeks
Population: Tabulations of the proportion of patients who achieved a hematologic normalization through end of study were performed for the ITT population. Exact 95% binomial confidence intervals were produced for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Percentage of Participants | 90 [68 to 99]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Percent of hematologic normalization = 90, 95% CI 2-sided [68 to 99]

9. Secondary Outcome: Percentage of Patients With Complete TMA Response
Description: The proportion of patients who achieved a Complete TMA Response from baseline through end of study with eculizumab was determined. Complete TMA Response was defined as Hematologic Normalization plus improvement in renal function (defined as (≥25% reduction from baseline in serum creatinine), which was sustained for two consecutive measurements over a period of at least four weeks.
Time Frame: Through End of Study, Median Exposure 156 Weeks
Population: Tabulations of the proportion of patients who achieved a complete TMA response from baseline through end of study were performed. For this endpoint, for any relevant proportions, exact binomial 95% confidence intervals were produced.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Percentage of Participants | 55 [32 to 77]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Percent of complete TMA response = 55, 95% CI 2-sided [32 to 77]

10. Secondary Outcome: TMA Intervention Rate
Description: TMA Intervention Rate (# PE/PI and # Dialysis Events/Patient/Day) in the eculizumab treatment period (from baseline through end of study) for PE/PI and (from the fifteenth day following the first eculizumab dose through end of study) for new dialysis events was compared with the TMA Intervention Rate during the pre-eculizumab treatment period.
Time Frame: Through End of Study, Median Exposure 156 Weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: #events/patient/day
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
#events/patient/day | 0.00 (0.02)
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.29

11. Secondary Outcome: Platelet Count Change From Baseline to 156 Weeks
Time Frame: From Baseline to 156 Weeks
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
10^9 cells/L | -3.68 [-25.15 to 17.79]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7307, ANOVA; [statistical method as in outcome 5, analysis 1]; LS mean change from baseline = -3.68, 95% CI 2-sided [-25.15 to 17.79]

12. Secondary Outcome: Percentage of Patients With Platelet Count Normalization
Description: Platelet count normalization was defined as the platelet count observed to be ≥150 x 10^9/L on at least two consecutive measurements which span a period of at least four weeks Not specified.
Time Frame: Through End of Study, Median Exposure 156 Weeks
Population: The tabulations of the proportion of patients who achieved platelet count normalization through end of study were performed for the ITT population. Exact binomial 95% confidence intervals were produced for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
Percentage of Participants | 90 [68 to 99]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Percent of platelet count normalization = 90, 95% CI 2-sided [68 to 99]

13. Secondary Outcome: Pharmacokinetics (PK) and Pharmacodynamics (PD); Minimum and Maximum Blood Concentration
Time Frame: Induction Phase for 4 weeks followed by Maintenance Phase starting on Week 5 through 26 weeks or longer.
Population: PK parameters Cmin and Cmax were estimated using a population PK model developed from the observed PK concentration data.
Measure: Mean (Standard Deviation); unit: micrograms/mil
Arm/Group | Eculizumab
Number analyzed (Participants) | 20
micrograms/mil
  max concentration during induction period | 161.47 (27.29)
  min concentration during induction period | 112.43 (16.98)
  max concentration during maintenance | 427.48 (67.54)
  min concentration during maintenance | 212.45 (53.75)

ADVERSE EVENTS:
Time Frame: Through end of study; Exposure to eculizumab in this study extended for a median of 156 weeks and ranged from 26 weeks to 182 weeks.
Description: At every visit, patients were asked a standard non-leading question to elicit any changes in their medical well-being including inquiry about any hospitalization, accidents, and new or changed concomitant medication regimens. AEs were also documented from any data collected (e.g. laboratory values, physical examination findings, ECG changes, etc.).
Arm/Group | Eculizumab
Serious Adverse Events (participants affected / at risk) | 13/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=20)
Pericardial effusion (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Medical device complication (General disorders) | 1
Amyloidosis (Immune system disorders) | 1
Transplant rejection (Immune system disorders) | 1
Bacteraemia (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Enterococcal infection (Infections and infestations) | 1
Gastroenteritis norovirus (Infections and infestations) | 1
Hepatitis E (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Post procedural infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Q fever (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Electrocardiogram T wave inversion (Investigations) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Catheter removal (Surgical and medical procedures) | 1
Limb operation (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 1
Vein disorder (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=20)
Abnormal clotting factor (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 7
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 3
Lymph node pain (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Microcytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 1
Deafness bilateral (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Motion sickness (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 4
Adrenal insufficiency (Endocrine disorders) | 1
Conjunctivitis (Eye disorders) | 1
Eye irritation Conjunctival haemorrhage (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Abdominal rigidity (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 10
Flatulence (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Gingival hyperplasia (Gastrointestinal disorders) | 1
Gingival ulceration (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Malaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Subileus (Gastrointestinal disorders) | 1
Tooth impacted (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 4
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 2
Extravasation (General disorders) | 1
Fatigue (General disorders) | 4
Hypothermia (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Infusion site swelling (General disorders) | 1
Injection site haematoma (General disorders) | 1
Localised oedema (General disorders) | 1
Malaise (General disorders) | 1
Medical device complication (General disorders) | 2
Medical device pain (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 6
Pain (General disorders) | 1
Polyp (General disorders) | 1
Pyrexia (General disorders) | 7
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatocellular injury (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 4
Seasonal allergy (Immune system disorders) | 1
Ateriovenous fistula site infection (Infections and infestations) | 1
BK virus infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Cytomegalovirus infection (Infections and infestations) | 1
Erythrasma (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 3
Infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 12
Otitis media (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 3
Vaginal infection (Infections and infestations) | 1
Viral pharyngitis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 2
Vulvovaginal candidiasis (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 4
Corneal abrasion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Foreign body (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 2
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Basophil count increased (Investigations) | 2
Blood creatine increased (Investigations) | 1
Blood creatinine increased (Investigations) | 4
Blood lactate dehydrogenase increased (Investigations) | 1
Blood parathyroid hormone increased (Investigations) | 2
Blood potassium increased (Investigations) | 1
Blood pressure abnormal (Investigations) | 1
Cardiac murmur (Investigations) | 2
Electrocardiogram T wave inversion (Investigations) | 1
Eosinophil count increased (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 1
Haptoglobin increased (Investigations) | 1
Low density lipoprotein increased (Investigations) | 1
Monocyte count increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Reticulocyte count increased (Investigations) | 1
Weight decreased (Investigations) | 3
White blood cell count increased (Investigations) | 1
White blood cells urine positive (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 2
Alkalosis (Metabolism and nutrition disorders) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Metabolism and nutrition disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haematoma (Nervous system disorders) | 1
Cerebral microangiopathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 11
Myoclonus (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Paresis (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Affective disorder (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 3
Breast swelling (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
Oedema genital (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Heat rash (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Rash macular (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
Arterial haemorrhage (Vascular disorders) | 1
Arterial occlusive disease (Vascular disorders) | 1
Haematoma (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 4
Orthostatic hypotension (Vascular disorders) | 2
Vein disorder (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participation in this multicenter study involved a commitment to publish the data from the study in a cooperative publication prior to release of study results on an individual basis.